CLINICAL TRIAL: NCT00180739
Title: Magnetic Resonance Guided Focused Ultrasound Surgery in the Treatment of Uterine Fibroids in Women Desiring Future Pregnancies
Brief Title: Safety Trial of Magnetic Resonance (MR) Guided Focused Ultrasound Surgery (FUS) in Women With Uterine Fibroids Wishing to Pursue Pregnancy in the Future
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment not possible worldwide
Sponsor: Imperial College London (Other)
Collaborators: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF004
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Uterine Fibroids; Pregnancy
Keywords: MR guided FUS; Uterine Fibroids; Fertility; Pregnancy
MeSH Terms: conditions — Leiomyoma

INTERVENTIONS:
Procedure: Magnetic Resonance Guided Focused Ultrasound

SUMMARY:
The study objective is to develop data for the safety of pregnancies after thermal ablation of uterine fibroids by MR guided Focused Ultrasound using the Ex Ablate 2000 system.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject with uterine fibroids, who desire pregnancy within 12 months and has the one of the following criteria: Women 20-40 age. Women age < 46 years old who plan to have egg donation. Women above 38 should test for normal ovarian function as judged by endocrinological evaluation.

If the couple has failed to conceive for more that 1 year, the woman should test for normal ovarian function as judged by endocrinological evaluation, and the male must have adequate sperm test.

Women undergoing fertility treatment or plan to have sperm donation.

* 2. Use or non use of non-steroidal treatments for excessive vaginal bleeding such as antifibrinolytic agents (e.g. Tranexamic acid) or non-steroidal anti-inflammatory drugs (e.g. Mefanamic Acid) has been maintained for the three months prior to the planned date of the study procedure and the patient has agreed to maintain this use or non-use through the 6-month follow-up period.
* 3. Clinically normal PAP smear within timing of National Guidelines in the country of the clinical site.
* 4. Able and willing to give consent and able to attend all study visits
* 5. Able to communicate sensations during the MRgFUS procedure
* 6. Having uterine fibroids that are device accessible (i.e., positioned in the uterus such that they can be accessed without being shielded by bowel or bone).
* 7. Tumor(s) are clearly visible on non-contrast MRI.
* 8. Largest fibroid 8 cm in diameter or 12 cm if receiving GnRH

Exclusion Criteria:

* 1. Patient is pregnant as confirmed by pregnancy test at time of screening
* 2. Uterine size >20 weeks as evaluated by US or MR.
* 3. Patients who are considered "high risk pregnancy" due to uterine factors (e.g. abnormal uterus, uterine scars, cerclage) except fibroids.
* 4. Patients with fibroid that is more than 50% sub-mucosal or with hysteroscopically resectable
* 5. Patients with adenomyosis
* 6. Patient is on dialysis
* 7. Hematocrit is < 25
* 8. Patient has hemolytic anemia
* 9. Patient has unstable cardiac status including: § Unstable angina pectoris on medication§ Documented myocardial infarction within 6 months of protocol entry§ Congestive heart failure requiring medication (other than diuretic)§ Currently taking anti-arrhythmic drugs§ Severe hypertension (diastolic BP>100 on medication)§ Presence of cardiac pacemaker
* 10. Patient has an ASA score of >2
* 11. Patient has severe cerebrovascular disease (multiple CVA or CVA within 6 months)
* 12. Patient is on anti-coagulation therapy or has an underlying bleeding disorder
* 13. Evidence of uterine pathology other than leiomyoma
* 14. Patient has an active pelvic infection or history of pelvic inflammatory disease
* 15. Patient has an undiagnosed pelvic mass outside the uterus.
* 16. Patient weight >110 kg
* 17. Subject with extensive abdominal scarring in an area of the abdomen directly anterior to the treatment area.
* 18. Subject with standard contraindications for MR imaging such as non-MRI compatable implanted metallic devices.
* 19. Known intolerance to the MRI contrast agent (e.g. Gadolinium or Magnevist).
* 20. Individuals who are not able or willing to tolerate the required prolonged stationary prone position during treatment (approximately 3 hours.)
* 21. Patient with an intrauterine contraceptive device anywhere in the treatment beam path.
* 22. Women who are breast feeding.
* 23. Five or more fibroids, bigger then 3cm diameter, each

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcomes in women who have received treatment with MRgFUS

SECONDARY OUTCOMES:
Efficacy of MRgFUS as judged by HRQOL questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Wady Gedroyc, Principal Investigator — St Mary's NHS Trust
Locations (1):
- St Mary's Hospital, London, United Kingdom

REFERENCES:
- [Background] Hindley J, Gedroyc WM, Regan L, Stewart E, Tempany C, Hynyen K, Mcdannold N, Inbar Y, Itzchak Y, Rabinovici J, Kim HS, Geschwind JF, Hesley G, Gostout B, Ehrenstein T, Hengst S, Sklair-Levy M, Shushan A, Jolesz F. MRI guidance of focused ultrasound therapy of uterine fibroids: early results. AJR Am J Roentgenol. 2004 Dec;183(6):1713-9. doi: 10.2214/ajr.183.6.01831713. PMID 15547216